CLINICAL TRIAL: NCT00182052
Title: Rosiglitazone (Avandia) vs. Placebo for Androgen Dependent Prostate Cancer: A Randomized Double-Blind, Placebo Controlled Phase III Study
Brief Title: Rosiglitazone (Avandia) vs. Placebo for Androgen Dependent Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Matthew R. Smith, MD, PhD, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 00-100; NCT00139412 (obsolete NCT alias)
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Adenocarcinoma of the Prostate; Prostate Cancer
Keywords: rosiglitazone; Avandia; androgen dependant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Drug: Rosiglitazone
- Group 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rosiglitazone — Given orally twice daily. Participants may continue study treatment as long as their disease does not progress and they don't experience any serious side effects.
  Other Names: Avandia
  Arms: Group 1
Other: Placebo — Given orally twice daily.
  Arms: Group 2

SUMMARY:
The purpose of this study it to learn the effects (good or bad) that rosiglitazone has on patients and their prostate cancer. This study is going to look at what effects rosiglitazone has on prostate specific antigen (PSA) levels.

DETAILED DESCRIPTION:
* Patients will be randomly assigned to initial treatment with either rosiglitazone or placebo orally twice daily, every day as long as there is no disease progression or serious side effects. Patients will be asked to complete a drug log to keep track of the medication.
* Before treatment begins the following tests will be performed: physical exam; bone scan; blood work (including PSA level test) and a urine sample.
* While on this study the following tests and procedures will be done once a month: review of side effects and routine blood tests (including PSA levels).
* While on this study the following tests and procedures will be done on months 2 and 4: review of side effects; routine blood tests (including PSA levels) and urine tests.
* If the patient's disease progressed the treatment code will be broken and if the patient was on placebo, they will have the option to begin taking rosiglitazone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Biochemical disease progression following local therapy defined as three rises in PSA with each PSA determination at least 4 weeks apart and each PSA value > or = 0.2ng/ml
* For men treated with radical prostatectomy, PSA > or = 2 ng/ml
* For men treated with primary radiation therapy or post-prostatectomy radiation therapy, PSA > or = 2 ng/ml and > 150% post-radiation nadir
* Not an appropriate candidate for salvage radiation therapy or salvage prostatectomy
* Baseline PSADT < 24 months
* CALGB performance status of 0,1 or 2

Exclusion Criteria:

* Metastatic disease
* Prior hormonal therapy for recurrent prostate cancer
* Prior chemotherapy for prostate cancer
* Current treatment with insulin or an oral hypoglycemic
* History of treatment with thiazolidinediones
* Radiation therapy within 6 months
* SGOT > 1.5 x ULN
* Fasting blood glucose < 60 mg/dl
* NYHA Class 3 or 4 cardiac status

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2000-09; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the activity of rosiglitazone by comparing changes in PSA doubling time between rosiglitazone-treated and placebo-treated men. | 3 years

SECONDARY OUTCOMES:
Evaluate time to PSA progression as a measure of the activity of rosiglitazone. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Smith, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Background] Smith MR, Manola J, Kaufman DS, George D, Oh WK, Mueller E, Slovin S, Spiegelman B, Small E, Kantoff PW. Rosiglitazone versus placebo for men with prostate carcinoma and a rising serum prostate-specific antigen level after radical prostatectomy and/or radiation therapy. Cancer. 2004 Oct 1;101(7):1569-74. doi: 10.1002/cncr.20493. PMID 15468186